CLINICAL TRIAL: NCT06560723
Title: Identifying and Managing Frailty in the Elderly in a Multiprofessional Health Home
Brief Title: Implementation of a Personalised Health Plan (PHP) on Patient Quality of Life Score at 2-year Follow-up
Acronym: FRAPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/0348/HP; 2023-A02358-37 (Other: French Minister)
Record Dates: First submitted 2024-07-18; First posted 2024-08-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Elderly, Frail
Keywords: identifying

STUDY DESIGN:
Intervention Model Description: The subjects included in this study will be described globally and then by group (experimental group and control group) using the usual parameters: mean, standard deviation, median, interquartile range, extreme values for quantitative variables; frequency and cumulative frequency (if relevant) for qualitative variables.
  For the primary endpoint, the variation in the SF-36 score between M0 and M24 will be calculated and compared between the two groups using Student's t test. This crude comparison will be supplemented by an adjusted comparison based on a linear regression model, taking into account sociodemographic and clinical characteristics deemed relevant to account for potential patient selection bias. These characteristics differ from one center to another, leading to a potential confounding bias, hence the proposed adjustment
Masking Description: Non Applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Interventional Arm (with PHP) (Other): The patient will have a standardized geriatric assessment carried out by a nurse in both Multiprofessional Health Home. This geriatric assessment will be used to draw up a summary with different objectives and priorities, which will then be discussed at a multi-professional consultation meeting in the month following the geriatric assessment. The first multi-professional consultation meeting (MCM) will present the summary of the geriatric assessment and discuss the care and assistance to be implemented in the Personalized Health Plan (PHP). The Personalized Health Plan will then be prepared and formalized by the nurse, in partnership with the other healthcare professionals involved in the Personalized Health Plan. It will be presented to and validated by the patient and his/her carer. The actions will then be implemented.
  Interventions: Diagnostic Test: Quality of life test
- Group 2 Control Arm (without PHP) (Other): In the control group, the attending physician will set up appropriate care for a patient identified as frail in a standard general medical care pathway, having been made aware of the patient's frailty at the time of inclusion. He or she will organize the patient's care, referring him or her to the appropriate specialists according to the difficulties identified at inclusion, and according to the patient's habits and network.
  Interventions: Diagnostic Test: Quality of life test

INTERVENTIONS:
Diagnostic Test: Quality of life test — The results of the various quality-of-life scores used to compile the study statistics (ADL, iADL, MMS, GDS, MNA, EPICES, SPPB, SF-36) will be provided to the doctor, but without any specific comments or recommendations, and then presented to the patient. Number of emergency room visits and hospitalization days, drug untake evalautions and thepareutic compliance (GIRERD score) will be also collected.

SUMMARY:
"Healthy ageing" is not limited to the absence of disease, but implies the "development and maintenance of the functional skills that enable the elderly to enjoy a state of well-being": (for example : the ability to walk, go out, engage in leisure activities, memorize...) It is interesting to study whether the implementation of a Personal Health Plan (PHP) in a Multiprofessional Health Home improves the quality of life of frail elderly people.

DETAILED DESCRIPTION:
"Healthy ageing" is not limited to the absence of disease, but implies the "development and maintenance of the functional skills that enable the elderly to enjoy a state of well-being": (for example : the ability to walk, go out, engage in leisure activities, memorize...) Between "good health" and "dependence", there is a precarious, reversible state of transition known as frailty. There are several simple tools for identifying frailty, such as the GFST (Gerontopole Frailty Screening Tool).

The Gerontopole Frailty Screening Tool and the Fatigue, Resistance, Ambulation, Illness, Loss of Weight questionnaire have proved more sensitive. The gold standard for diagnosing and assessing frailty is a comprehensive geriatric assessment based on the multidimensional model of the Standardized Geriatric Assessment (SGA). Its aim is to identify all the medical, functional, psychological and social problems that may affect a frail elderly patient, in order to set up a long-term follow-up project, taking into account the patient's needs.

It is interesting to study whether the implementation of a Personal Health Plan in a Multiprofessional Health Home improves the quality of life of frail elderly people.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 70 years
* Autonomous patient (ADL ≥ 5)
* Patient identified as frail according to the Gérontopôle de Toulouse GFST grid
* Patient whose primary care physician is in the MSPs of Charleval or Romilly sur Andelle for the intervention group, and in the MSPs of Gaillon and Pont de l'Arche for the control group.
* Patient living at home or in an RPA
* Understanding of the French language
* Patient having read and understood the information letter and signed the consent form
* Affiliation with a social security scheme

Exclusion Criteria:

* Hospital geriatric follow-up
* Geriatric assessment already carried out
* Person deprived of liberty by an administrative or judicial decision, or placed under court protection / sub-guardianship or curatorship
* History of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol, or from giving informed consent.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of implementing a personalized healthcare plan (PPS) on patient quality of life at M24 | 2 years
  change in Study short Form -36 (SF-36) quality-of-life score between Inclusion (M0) and 2-year follow-up (M24). The SF-36 consists of 36 questions to assess quality of life related to general health. Each item is scored on a scale from 0 to 100, 0 and 100 representing the lowest and highest possible scores

SECONDARY OUTCOMES:
Patient quality of life at M6 and M12 | 1 year
  Patient quality of life, measured by SF-36 score, at M0, M6 and M12. The SF-36 consists of 36 questions to assess quality of life related to general health. Each item is scored on a scale from 0 to 100, 0 and 100 representing the lowest and highest possible scores
Emergency room visits and hospitalizations at M6, M12 and M24 | 2 years
  Number of emergency room visits and hospital days at M6, M12 and M24
Drug intake at M6, M12 and M24 | 2 years
  Number of medications taken at M6, M12 and M24
Therapeutic compliance at M6, M12 and M24 | 2 years
  Therapeutic compliance, measured by GIRERD questionnaire score at M0, M6, M12 and M24. The GIRERD Questionnaire is a Self-questionnaire to estimate the level of compliance, namely whether the treatment is taken regularly and as prescribed. All responses are rated as "yes" or "no". One "yes" is equivalent to one point. Score = 0: Good compliance. Score = 1 or 2: Minor compliance issue. Score 3: Poor compliance.
Patient autonomy at M6, M12 and M24. | 2 years
  Autonomy, measured by ADL score at M0, M6, M12 and M24.
  - Activities of Daily Living (ADL) score helps to know if a person needs human help in the basic gestures of everyday life. A score of 6 determines the maximum level of autonomy.
Falls and patient mobility at M6, M12 and M24 | 2 years
  Assessment of mobility measured by number of falls and SPPB (Short Physical Performance Battery) score at M0, M6, M12 and M24. The SPPB (Short Physical Performance Battery) is the sum of scores on three criteria: the balance test, the walking speed test and the chair lift test. This test is used to assess the physical performance of an individual. The addition of scores from all tests gives an overall performance score. A score below 8 is an indicator of risk for sarcopenia (or age-related muscular dystrophy)
Patient nutritional status at M6, M12 and M24 | 2 years
  Nutritional status, measured by MNA test score at M0, M6, M12 and M24
Patient's cognitive status at M6, M12 and M24 | 2 years
  Cognitive status, measured by MMS score at M0, M6, M12 and M24. The Mini-Mental State Examination allows for a cognitive assessment of the patient. A score at the end of the test less than or equal to 24 points can evoke an altered state of consciousness and direct.
Patient's emotional state at M6, M12 and M24 | 2 years
  Emotional state, measured by the 15-question GDS questionnaire score at M0, M6, M12 and M24. Geriatric Depression ScaleScore is used to identify depressive symptoms in elderly people. 0-5: normal; Score between 5 and 9: indicates a high probability of depression; Score 10 and above: almost always indicates depression.
Patient's social fragility at M6, M12 and M24 | 2 years
  Social fragility, measured by the EPICES questionnaire score, at M0, M6, M12 and M24. The EPICES score (Evaluation of Precariousness and Health Inequalities in Examination Centers Health) is an individual indicator of poverty. The score is between 0 (absence of precariousness) and 100 (maximum of precariousness).
Patient autonomy at M6, M12 and M24. | 2 years
  Autonomy, measured by iADL score at M0, M6, M12 and M24.
  - Instrumental Activities of Daily Living (iADL) score shows the level of autonomy of the patient: a maximum score of 8 represents a maximum autonomy and the more the score decreases, the more the level of autonomy decreases. This test is very fast to use and allows you to identify some dependencies.

OTHER OUTCOMES:
Cost/Utility analysis at M12 and M24 | 2 years
  All direct medical and non-medical costs will be considered from inclusion up to 24 months, and will be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Lucille PELLERIN, Dr, Study Chair — Rouen University Department of General Medicine